CLINICAL TRIAL: NCT03474887
Title: Digital Online Consultations - Effects on Antibiotic Prescribing and Health Care Utilization in Primary Care
Acronym: DOCACUP
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Doctrin (Unknown); Capio Group (Other); Capio Go (Unknown); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/948
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Sore Throat; Dysuria; Cough; Common Cold; Influenza
Keywords: Telemedicine; Remote consultation; Mobile health; Telehealth; mhealth; eVisits; eConsultation; ehealth
MeSH Terms: conditions — Pharyngitis; Dysuria; Cough; Common Cold; Influenza, Human | interventions — Office Visits

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- DIGI-Throat: Patients choosing to seek primary care through an online consultation with chief complaint sore throat.
  Interventions: Other: Online Consultation
- DIGI-Resp: Patients choosing to seek primary care through an online consultation with chief complaint cough/common cold/influenza.
  Interventions: Other: Online Consultation
- DIGI-Dysuria: Patients choosing to seek primary care through an online consultation with chief complaint dysuria.
  Interventions: Other: Online Consultation
- PHYSI-Throat+CONTROL-Throat: Patients choosing to seek primary care through physical consultation with chief complaint sore throat.
  + Patients seeking primary care prior to implementation of online consultations, with a chief complaint of sore throat.
  Interventions: Other: Physical Consultation
- PHYSI-Resp+CONTROL-Resp: Patients choosing to seek primary care through physical consultation with chief complaint cough/common cold/influenza.
  + Patients seeking primary care prior to implementation of online consultations, with a chief complaint of cough/common cold/influenza.
  Interventions: Other: Physical Consultation
- PHYSI-Dysuria+CONTROL-Dysuria: Patients choosing to seek primary care through physical consultation with chief complaint dysuria
  + Patients seeking primary care prior to implementation of online consultations, with a chief complaint of dysuria.
  Interventions: Other: Physical Consultation

INTERVENTIONS:
Other: Physical Consultation — Regular physician consultation at the primary care clinic.
  Other Names: Office Visit
  Groups: PHYSI-Dysuria+CONTROL-Dysuria; PHYSI-Resp+CONTROL-Resp; PHYSI-Throat+CONTROL-Throat
Other: Online Consultation — An online platform for communicating with a physician digitally. Patients answer a series of algorithm-based questions after specifying chief complaint, after which contact is established with a physician who can communicate through short messages. The physician can then order labs, prescribe relevant medication or book the patient for a physical consultation if need be.
  Other Names: eVisit; Capio Go; Lakarbesok online
  Groups: DIGI-Dysuria; DIGI-Resp; DIGI-Throat

SUMMARY:
BACKGROUND/SIGNIFICANCE: With developments in mobile health and the abundance of smartphones, online consultations have emerged as a popular form of primary care in Sweden. Controversy exists regarding diagnostic accuracy, appropriate prescription of antibiotics, and effects on care-seeking patient behavior following implementation of online consultations. As empirical research is lacking, the investigators seek to evaluate online primary care consultations compared to physical consultations with regards to non-inferiority of antibiotic prescription for chief complaint of sore throat.

METHODS: Medical record data is used to identify patients with a chief complaint of sore throat, cough/common cold/influenza, or dysuria after choosing online (DIGI) or physical (PHYSI) consultations. A cohort of patients with similar chief complaints prior to implementation of online consultations was used as a control group (CONTROL). Prospective data from local registries and medical records was gathered 14 days the consultation. The primary outcome was rate of antibiotic prescription after sore throat. Secondary outcomes included patient revisits (including hospital admissions), patient satisfaction, time to physician contact, registered diagnosis, and documentation or Centor Criteria and Urinary Tract Infection (UTI)-Criteria.

SIGNIFICANCE: Results will shed light on whether antibiotic prescription differs significantly between digital and physical primary care consultations. Hypotheses may also be generated as to how patients seek care in light of improved availability in a tax-sponsored healthcare system.

DETAILED DESCRIPTION:
Due to limited recruitment of PHYSI and CONTROL patients, these cohorts will be combined into a single physical cohort to provide adequate power for analysis as per predefined required sample size.

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking care at primary healthcare provider (Capio in Skåne or Capio Go)
* Patient who according to medical record presents with sore throat, cough/common cold/influenza, or dysuria

Exclusion Criteria:

* Patient who according to medical record presents with main symptom other than sore throat, cough/common cold/influenza, or dysuria.
* Patient under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators seek to emulate a primary care cohort in order to make the evaluation of physical and online consultations comparable.
Sampling Method: Non-Probability Sample
Enrollment: 4057 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Antibiotics Prescription After Sore Throat | 24 hours
  Proportion of patients prescribed an antibiotics (as documented in medical records) in conjunction with their initial visit with chief complaint sore throat.

SECONDARY OUTCOMES:
Antibiotics Prescription After Cough/Common Cold/Influenza | 24 hours
  Proportion of patients prescribed an antibiotics (as documented in medical records) in conjunction with their initial visit with chief complaint cough/common cold/influenza.
Antibiotics Prescription After Dysuria | 24 hours
  Proportion of patients prescribed an antibiotics (as documented in medical records) in conjunction with their initial visit with chief complaint dysuria.
Patient Revisits | 14 days
  Number of healthcare-system visits following initial consultation (as documented in local registries). Includes outpatient as well as inpatient visits.
Type of Antibiotic Prescribed | 24 hours
  ATC-codes of antibiotics prescribed in conjunction with the initial consultation.
Registered Diagnosis | 24 hours
  Diagnosis registered in with medical journal in conjunction with with initial consultation.
Patient Satisfaction | 24 hours
  Average scores documented on a 3 question survey, if documented.
Time to Physician Contact | 14 days
  DIGI: Time from patient log-in on the online platform to first speech-bubble from the physician.
  PHYSI and CONTROL: Time from registered telephone contact to registered physician contact.
Centor Criteria Documentation | 24 hours
  Proportion of patients where Centor Criteria are fully documented in the medical record in conjunction with the initial consultation.
  Centor criteria: Tonsillar redness/exudates, Tender anterior cervical adenopathy, fever over 38,5° C, absence of cough.
UTI Criteria Documentation | 24 hours
  Proportion of patients where urinary tract infection criteria are fully documented in the medical record in conjunction with the initial consultation.
  UTI Criteria: increased pain, frequency, urgency. Lack of vaginal symptoms, fever or flank pain.
Ordering of labs for sore throat | 24 hours
  Defined as "StrepA" quick-test for group A Streptococcus (GAS)-tonsillitis, including outcome
Ordering of labs for dysuria | 24 hours
  Defined as urinalysis, including outcomes of leukocytes and nitrate

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundkvist, Professor, Study Chair — CPF, Department of Clinical Sciences, Malmö
Locations (1):
- Capio Go, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Entezarjou A, Sjobeck M, Midlov P, Nymberg VM, Vigren L, Labaf A, Jakobsson U, Calling S. Health care utilization following "digi-physical" assessment compared to physical assessment for infectious symptoms in primary care. BMC Prim Care. 2022 Jan 12;23:4. doi: 10.1186/s12875-021-01618-2. eCollection 2022. PMID 35036998
- [Derived] Entezarjou A, Calling S, Bhattacharyya T, Milos Nymberg V, Vigren L, Labaf A, Jakobsson U, Midlov P. Antibiotic Prescription Rates After eVisits Versus Office Visits in Primary Care: Observational Study. JMIR Med Inform. 2021 Mar 15;9(3):e25473. doi: 10.2196/25473. PMID 33720032